CLINICAL TRIAL: NCT02995213
Title: Quantification of UE Use and Effects of Feedback in the Home Setting
Acronym: OPTASpr2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Maureen Whitford, Assistant Professor, Cleveland State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2016-84
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Feedback Intervention (Experimental)
  Interventions: Behavioral: Accelerometer based feedback about paretic arm use

INTERVENTIONS:
Behavioral: Accelerometer based feedback about paretic arm use

SUMMARY:
The investigators are proposing a pilot study, the purpose of which is to use accelerometers to quantify UE use (1 and two hand use) in people post-stroke from which the investigators will develop use-based feedback to improve recovery in the home setting. The objectives of this pilot study are to:

i.) determine the feasibility of using accelerometers to quantify amount of UE use in the home setting in individuals chronic post-stroke,

ii.) quantify and compare the unilateral activity of the weaker (paretic) versus stronger (non-paretic) UEs, and

iii.) assess the effect of a 7 sessions of in-home accelerometer used-based feedback on unilateral and bilateral UE use.

iv.) assess kinematic, kinetic, and EMG data during UE movements unilaterally and bilaterally in subjects post-chronic stroke pre and post feedback.

ELIGIBILITY:
Inclusion Criteria:

* Subjects post-stroke
* chronic post ischemic or hemorrhagic cortical or subcortical stroke
* 25 - 100 years old
* upper extremity impairment
* Subjects will need to be able to flex their paretic shoulder and their elbow > 40° without assist
* able to follow 2-step commands
* community dwelling with or without assistance
* intact superficial light touch sensation in both upper extremities
* must also have some movement in both arms

Exclusion Criteria:

* can't currently have another neuromuscular disorders such as spinal cord injury, traumatic brain injury, Parkinson disease or multiple sclerosis
* no upper extremity injury within the last 3 months

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Accelerometer based paretic arm amount of use | 3 week period

IPD SHARING:
Plan to Share IPD: No